CLINICAL TRIAL: NCT05811559
Title: Investigation of the Relationship Between Sensory Processing and Potential Impact Factors in Elderly Adults Receiving Hip Fracture Surgery for Falling
Brief Title: Investigation of Sensory Processing Patterns of Elderly Individuals Who Have Had Hip Fracture Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Sena Erarslan, Principal Investigator, Atlas University
Other Study IDs: SErarslan2023-1
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Sensory Disorder; Sensory Processing Disorder; Hip Fractures; Fall Injury; Falling; Sensitivity; Elderly
MeSH Terms: conditions — Sensation Disorders; Hip Fractures; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to evaluate the sensory processing processes of elderly adults who have undergone fall-related hip fracture surgery in the last 6 months, according to different patterns, and to examine the relationship between physical performance, fall risk, fear of falling, and depression parameters that may be related to sensory processing.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Being able to stand independently for 30 seconds
* Being able to walk 3 m independently (with an assistive device if necessary)
* Getting a score of 24 or more on the Mini Mental Test

Exclusion Criteria:

* Hip fracture patients receiving medical treatment for pathological hip fractures, polytrauma, traffic accidents, bone tumors
* Having a history of diseases that may directly affect the evaluation process (neurological diseases such as Parkinson's, Alzheimer's and cancer)
* Having vision and hearing loss
* Having a psychiatric illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adult individuals who have suffered a fall and therefore undergo hip fracture surgery.
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Adult Sensory Processing Scale | 20 minutes
  The Adult Sensory Processing Scale is a self-report tool developed to measure the response given to stimuli from different sensory systems in adults, sensitive to individual differences. Scale; evaluates different behavioral responses (overreaction, underreaction and sensory seeking) in five different sensory systems, namely tactile, proprioceptive, vestibular, visual and auditory, which are indicators of sensory processing difficulties. The scale consists of 11 factors and 48 items in total. All items are rated on a 5-point Likert scale as never = 1, rarely = 2, sometimes = 3, often = 4, and always = 5. While calculating the scale, the scores obtained from each factor are graded in 3 different categories: "typical range", "possible difficulty" and "exact difficulty".
Short Physical Performance Battery | 25 minutes
  Short Physical Performance Battery, consists of 3 performance-based tests that evaluate standing balance, walking speed and sitting balance, and which are simple and faster to use clinically than other fall risk tools. The performance time of each performed task is recorded with a stopwatch. Each performance test is scored between 1-4. If the task given in the test cannot be completed, 0 points are recorded. A total score in the range of 0-12 is obtained by summing the scores of all performance areas. High scores mean good performance .
Timed Up and Go Test | 5 minutes
  It is a practical and reliable measurement tool that evaluates fall risk and mobility in elderly individuals. During the test, the participant is sitting in a standard chair with a seat height of approximately 46 cm. With the therapist's start command, the participant is asked to get up from the chair, walk up to the marked distance of 3 meters, turn back and sit back in the chair. To measure performance, the elapsed time is recorded in seconds.
Falls Efficacy Scale | 10 minutes
  Scale; It aims to evaluate the self-confidence of the individual in the realization of 10 activities that are relatively safe from daily life activities without falling. The individual is asked to give a score between 1 and 10 on a numerical scale for each activity. 1 point means I don't trust at all, 10 points means I trust very much and all points are added to get the total score of the test. The total score that can be obtained from the scale is in the range of 10-100. An increase in the score indicates the presence of less safe behaviors related to falling.
Geriatric Depression Scale | 15 minutes
  The scale was specifically designed by Yesavage et al. The easy-to-understand, self-reported 30-item scale includes questions about affective changes, negative attitudes about the past, present and future, and withdrawal from life. By summing all the items, a total score ranging from 0-30 is obtained. It is reported that the risk of depression is high for older adults who score 14 points or more.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided